CLINICAL TRIAL: NCT02175641
Title: Peer-Led Healthy Lifestyle Program in Supportive Housing Agencies
Brief Title: Peer-Led Healthy Lifestyle Program in Supportive Housing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Leopoldo J. Cabassa, Associate Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAN5207; 1R01MH104574-01 (NIH)
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Results first posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Obesity
Keywords: Healthy lifestyle Intervention; Serious Mental Illness; Effectiveness trial; Supportive housing; Racial and Ethnic Health Disparities
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peer-led Group Lifestyle Balance (Experimental): Group-based behavioral healthy lifestyle program
  Interventions: Behavioral: Peer-Led Group Lifestyle Balance; Behavioral: Usual Care Services
- Usual Care Services (Active Comparator): Usual wellness and health care services offered to clients at the two supportive housing agencies.
  Interventions: Behavioral: Usual Care Services

INTERVENTIONS:
Behavioral: Peer-Led Group Lifestyle Balance — The intervention follows the Group Lifestyle Balance curriculum derived from the Diabetes Prevention Program and The intervention will be delivered by trained peer-specialists employed at the supportive housing agencies and supervised by the study team. Peer GLB is a 12-month group intervention that focuses helping people lose weight by improving people's diet and increasing their physical activity and consists of weekly core group sessions (3 mo.), bi-monthly transitional group sessions (3 mo.), and maintenance monthly sessions (6 mo.).
  Arms: Peer-led Group Lifestyle Balance
Behavioral: Usual Care Services — The usual care condition encompasses the regular services offered at supportive housing agencies to help clients with their physical health and wellness.

SUMMARY:
This goal of this randomized controlled effectiveness trial is to compare the effectiveness of a peer-led health lifestyle intervention (Peer GLB) versus usual care services in supportive housing agencies in New York City and Philadelphia serving diverse clients with serious mental illness who are overweight or obese. The intervention follows the Group Lifestyle Balance curriculum derived from the Diabetes Prevention Program and that has been shown to help people achieve clinically significant weight loss (equal to or greater than 5% weight loss of initial weight). The intervention will be delivered by trained peer-specialists employed at the supportive housing agencies and supervised by the study team. Peer GLB is a 12-month group intervention that focuses helping people lose weight by improving people's diet and increasing their physical activity and consists of weekly core group sessions (3 mo.), bi-monthly transitional group sessions (3 mo.), and maintenance monthly sessions (6 mo.).

We plan to enroll 300 clients with serious mental illness who are overweight/obese (BMI equal to or greater than 25) from our two supportive housing agencies. Clients will be randomized to either the Peer-led healthy lifestyle intervention or usual care conditions. The primary outcome for this study is achieving clinically significant weight loss (equal to or greater than 5% weight loss from baseline weight) at 12 and 18 months post randomization. The secondary outcomes for this study include overall reductions in weight, waist circumference, blood pressure, and improvements in physical activity, self-efficacy, recovery and health-related quality of life. Repeated assessments will be at baseline, 6, 12 and 18 month post randomization.

Primary Hypothesis: Peer GLB participants will have a higher proportion of persons achieving clinically significant weight loss (equal to or greater than 5% weight loss) at 12 and 18 months than UC participants.

Secondary Hypothesis: At 6, 12, and 18 months post-randomization, there will be significant reductions in average weight, waist circumference, blood pressure, and significant improvements in physical activity, self-efficacy, recovery, and health-related quality of life in Peer GLB compared to UC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female,18 years of age or older, of any race/ethnicity, who are English and/or Spanish speakers.
* Chart diagnosis of a serious mental illness (SMI; e.g., schizophrenia, bipolar disorder, schizoaffective disorders, major depression).
* Overweight/obese as determined by a Body Mass Index (BMI) equal to or greater than 25 (kg/m2) at the time of recruitment.
* Able and willing to give informed consent and participate in the intervention.
* Received a medical clearance from a primary care or medical provider to participate in light-to-moderate physical activity (e.g., 150 minutes a week of brisk walking).

Exclusion Criteria:

* Need for detoxification services at the time of recruitment.
* Pose a danger to self or others at the time of recruitment.
* Have medical conditions that contraindicate their participation in a healthy lifestyle program focusing on weight loss and physical activity, such as active cancer treatment, liver failure, history of anorexia nervosa, cardiovascular event [e.g., unstable angina, myocardial infraction] within the past 6 months, untreated exercise- induced asthma, walking limitations preventing participation in exercise, and pregnant or planning a pregnancy during study period.
* Fail a capacity-to-consent questionnaire.
* Cognitive impairment as detected by the Mini-Cog Examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo J Cabassa, Ph. D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cabassa LJ, Stefancic A, O'Hara K, El-Bassel N, Lewis-Fernandez R, Luchsinger JA, Gates L, Younge R, Wall M, Weinstein L, Palinkas LA. Peer-led healthy lifestyle program in supportive housing: study protocol for a randomized controlled trial. Trials. 2015 Sep 2;16:388. doi: 10.1186/s13063-015-0902-z. PMID 26329472
- [Derived] Tuda D, Stefancic A, Hawes M, Wang X, Guo S, Cabassa LJ. Correlates of Attendance in a Peer-Led Healthy Lifestyle Intervention for People with Serious Mental Illness Living in Supportive Housing. Community Ment Health J. 2022 May;58(4):761-769. doi: 10.1007/s10597-021-00881-y. Epub 2021 Aug 20. PMID 34417635
- [Derived] Stefancic A, Bochicchio L, Tuda D, Harris Y, DeSomma K, Cabassa LJ. Strategies and Lessons Learned for Supporting and Supervising Peer Specialists. Psychiatr Serv. 2021 May 1;72(5):606-609. doi: 10.1176/appi.ps.202000515. Epub 2021 Mar 4. PMID 33657843
- [Derived] Stefancic A, Bochicchio L, Tuda D, Gurdak K, Cabassa LJ. Participant Experiences With a Peer-Led Healthy Lifestyle Intervention for People With Serious Mental Illness. Psychiatr Serv. 2021 May 1;72(5):530-538. doi: 10.1176/appi.ps.202000311. Epub 2021 Mar 4. PMID 33657839
- [Derived] Stefancic A, Bochicchio L, Svehaug K, Alvi T, Cabassa LJ. "We Die 25 Years Sooner:" Addressing Physical Health Among Persons with Serious Mental Illness in Supportive Housing. Community Ment Health J. 2021 Aug;57(6):1195-1207. doi: 10.1007/s10597-020-00752-y. Epub 2021 Jan 1. PMID 33385266
- [Derived] Cabassa LJ, Stefancic A, Lewis-Fernandez R, Luchsinger J, Weinstein LC, Guo S, Palinkas L, Bochicchio L, Wang X, O'Hara K, Blady M, Simiriglia C, Medina McCurdy M. Main Outcomes of a Peer-Led Healthy Lifestyle Intervention for People With Serious Mental Illness in Supportive Housing. Psychiatr Serv. 2021 May 1;72(5):555-562. doi: 10.1176/appi.ps.202000304. Epub 2020 Dec 18. PMID 33334158

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peer-led Group Lifestyle Balance | Usual Care Services
Started | 157 | 157
6-month Follow up | 144 | 149
12-month Follow up | 129 | 136
18-month Follow up | 122 | 130
Completed | 122 | 130
Not Completed | 35 | 27
Not completed — Death | 3 | 4
Not completed — Lost to Follow-up | 4 | 4
Not completed — Withdrawal by Subject | 7 | 4
Not completed — Discharged from Supportive Housing Agenc | 13 | 15
Not completed — Developed Contraindicated Condition | 8 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer-led Group Lifestyle Balance | Usual Care Services | Total
Number analyzed (Participants) | 157 | 157 | 314
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.50 (11.56) | 48.81 (11.60) | 48.65 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 66 | 133
  Male | 90 | 91 | 181
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 28 | 29 | 57
  Non-Hispanic Black | 104 | 77 | 181
  Hispanic | 13 | 26 | 39
  Other | 12 | 25 | 37
Weight [Mean (Standard Deviation); unit: Pounds] | 225.75 (58.07) | 211.84 (48.83) | 218.79 (54.01)

OUTCOME MEASURES:

1. Primary Outcome: Clinically Significant Weight Loss
Description: Percentage of participants that achieve equal to or greater than 5% weight loss in lb from baseline at 12 and 18th months
Time Frame: Baseline to 18 Months
Population: Participants enrolled in the trial and randomized to either Peer-led Group Lifestyle Balance or Usual Care Services
Measure: Count of Participants; unit: Participants
Arm/Group | Peer-led Group Lifestyle Balance | Usual Care Services
Number analyzed (Participants) | 122 | 130
Participants | 39 | 40
Statistical Analysis 1: Comparison: Peer-led Group Lifestyle Balance vs Usual Care Services; Test type: Other — Generalized linear mixed-effects models with a logistic link; p > 0.05, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.62 to 1.84]

2. Secondary Outcome: Overall Reduction in Weight in lb From Baseline to 6, 12 and 18 Months
Description: Weight (in pounds) was measured by a trained research assistant with a calibrated digital scale (participants wore indoor clothing without shoes).
Time Frame: At study endpoint (18 months).
Population: Participants enrolled in the trial and randomized to either Peer-led Group Lifestyle Balance or Usual Care Services. Results presented are weight at the study endpoint (18-months).
Measure: Mean (Standard Deviation); unit: lb
Arm/Group | Peer-led Group Lifestyle Balance | Usual Care Services
Number analyzed (Participants) | 122 | 130
lb | 226.04 (62.81) | 209.51 (50.41)
Statistical Analysis 1: Comparison: Peer-led Group Lifestyle Balance vs Usual Care Services; Test type: Other — Mixed effect models controlling for study site; p = 0.804, Mixed Models Analysis; Time by treatment interaction coefficien = 0.15, Standard Error of Mean 0.59

3. Secondary Outcome: Overall Reduction in Waist Circumference Measures to the Nearest cm From Baseline to 6, 12 and 18 Months
Description: Waist circumference measured by a trained research assistant to the nearest 0.1 cm with an anthropometric tape, in a horizontal plane 1 cm above the navel in light indoor clothing.
Time Frame: At study endpoint (18 months).
Population: Participants enrolled in the trial and randomized to either Peer-led Group Lifestyle Balance or Usual Care Services.
Measure: Mean (Standard Deviation); unit: centimeters (CM)
Arm/Group | Peer-led Group Lifestyle Balance | Usual Care Services
Number analyzed (Participants) | 121 | 128
centimeters (CM) | 114.61 (18.84) | 110.38 (16.91)
Statistical Analysis 1: Comparison: Peer-led Group Lifestyle Balance vs Usual Care Services; Test type: Other; p = 0.91, Mixed Models Analysis; Time*treatment interaction coefficient = 0.05, Standard Error of Mean 0.09

4. Secondary Outcome: Overall Reductions in Systolic Blood Pressure From Baseline, 6, 12 and 18 Months
Description: Blood pressure assessed on the right arm of participants after they rest quietly in a seated position for at least 5 minutes, using a validated automated sphygmomanometer.
Time Frame: At study endpoint (18 months).
Population: Participants enrolled in the trial and randomized to either Peer-led Group Lifestyle Balance or Usual Care Services.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Peer-led Group Lifestyle Balance | Usual Care Services
Number analyzed (Participants) | 113 | 127
Millimeters of mercury (mmHg) | 129.52 (17.70) | 128.28 (19.13)
Statistical Analysis 1: Comparison: Peer-led Group Lifestyle Balance vs Usual Care Services; Test type: Other — Mixed effect models controlling for study site; p = 0.64, Mixed Models Analysis; time*treatment interaction coefficient = -0.34, Standard Error of Mean 0.74

5. Secondary Outcome: Self-Efficacy for Exercise
Description: Self-efficacy for exercise was measured with a three-item scale assessing a person's confidence that they can engage in physical activity. The scores from this scale range from 1 to 10 with higher scores indicating higher self-efficacy.
Time Frame: At study endpoint (18 months).
Population: Participants enrolled in the trial and randomized to either Peer-led Group Lifestyle Balance or Usual Care Services.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Peer-led Group Lifestyle Balance | Usual Care Services
Number analyzed (Participants) | 120 | 130
Score on a scale | 6.73 (2.58) | 6.89 (2.32)
Statistical Analysis 1: Comparison: Peer-led Group Lifestyle Balance vs Usual Care Services; Test type: Other — Mixed effect models controlling for study site; p = 0.38, Mixed Models Analysis; Time*treatment interaction coefficient = 0.08, Standard Error of Mean 0.09

6. Secondary Outcome: Change From Baseline in Recovery Using the Recovery Assessment Scale (RAS).
Description: The Recovery Assessment Scale is a 24-item measure that captures different aspects of recovery and produces a total recovery score ranging from 1 to 5 with higher scores indicating higher recovery.
Time Frame: At study endpoint (18 months).
Population: Participants enrolled in the trial and randomized to either Peer-led Group Lifestyle Balance or Usual Care Services.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer-led Group Lifestyle Balance | Usual Care Services
Number analyzed (Participants) | 120 | 129
score on a scale | 4.26 (0.64) | 4.26 (0.57)
Statistical Analysis 1: Comparison: Peer-led Group Lifestyle Balance vs Usual Care Services; Test type: Other — Mixed effect models controlling for study site; p = 0.39, Mixed Models Analysis; Time*treatment interaction coefficient = 0.02, Standard Error of Mean 0.02

7. Secondary Outcome: Health-related Quality of Life
Description: The 12-Item Short-Form Health Survey (SF-12) was used to capture participants health-related quality of life. The Physical Composite Score derived from the SF-12 is an indicator of health-related quality of life with scores that range from 0 to 100 with higher scores indicating higher health-related quality of life.
Time Frame: At study endpoint (18-months).
Population: Participants enrolled in the trial and randomized to either Peer-led Group Lifestyle Balance or Usual Care Services.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer-led Group Lifestyle Balance | Usual Care Services
Number analyzed (Participants) | 118 | 129
score on a scale | 44.81 (10.36) | 45.71 (10.26)
Statistical Analysis 1: Comparison: Peer-led Group Lifestyle Balance vs Usual Care Services; Test type: Other — Mixed effect models controlling for study site; p = 0.52, Mixed Models Analysis; Time*treatment interaction coefficient = 0.23, Standard Error of Mean 0.37

8. Secondary Outcome: 6-Minutes Walking Test
Description: The 6-minutes Walking Test is an objective measure of functional exercise capacity that captures the distance (in meters) that participants walk at a normal pace along a flat and straight course for 6 minutes.
Time Frame: At study endpoint (18-months).
Population: Participants enrolled in the trial and randomized to either Peer-led Group Lifestyle Balance or Usual Care Services.
Measure: Mean (Standard Error); unit: meters
Arm/Group | Peer-led Group Lifestyle Balance | Usual Care Services
Number analyzed (Participants) | 117 | 126
meters | 315.83 (95.97) | 318.16 (93.38)
Statistical Analysis 1: Comparison: Peer-led Group Lifestyle Balance vs Usual Care Services; Test type: Other — Mixed effect models controlling for study site; p = 0.24, Mixed Models Analysis; Time*treatment interaction coefficient = 3.83, Standard Error of Mean 3.28

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Peer-led Group Lifestyle Balance | Usual Care Services
All-Cause Mortality (participants affected / at risk) | 3/157 | 4/157
Serious Adverse Events (participants affected / at risk) | 21/157 | 21/157
Other Adverse Events (participants affected / at risk) | 0/157 | 0/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peer-led Group Lifestyle Balance (N=157) | Usual Care Services (N=157)
Acquired Immunodeficiency Syndrome (Immune system disorders) | 1 | 0
Kidney Infection (Renal and urinary disorders) | 0 | 1
Cystitis (Renal and urinary disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 1
Stroke (Vascular disorders) | 0 | 3
Transient Ischemic Attack (Vascular disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 2 | 0 — Resulted in Death
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Wound Infection (Infections and infestations) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound Decomposition (Injury, poisoning and procedural complications) | 0 | 1
Stab Wound (Injury, poisoning and procedural complications) | 1 | 0
Foreign Body (Injury, poisoning and procedural complications) | 1 | 0
Drug Toxicity (Injury, poisoning and procedural complications) | 1 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Dyspnoaea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstrucive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Resulted in Death
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hernia Repair (Surgical and medical procedures) | 0 | 1
Cyst Removal (Surgical and medical procedures) | 1 | 0
Adverse Drug Reaction (General disorders) | 2 | 0
Death NOS (General disorders) | 2 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Brain Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Liver Disorder (Hepatobiliary disorders) | 0 | 1 — Resulted in Death

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT02175641/Prot_SAP_000.pdf